

# TRIAL STATISTICAL ANALYSIS PLAN MODULE A (BI 754091 + BI 754111)

c38788170-01

**BI Trial No.:** 1381.9

**Title:** An open-label, Phase II trial evaluating the safety and efficacy of

BI 754111 in combination with BI 754091 in in PD-(L)1 naïve and

PD-(L)1 pretreated patient populations with advanced and/or

metastatic solid tumours who have had at least one line of systemic

therapy

Investigational Product(s):

BI 754091 (anti-PD-1)

BI 754111 (anti-LAG-3)

Responsible trial statistician(s):

Phone:

Date of statistical

04 MAY 2022 SIGNED

analysis plan:

Version: Final


**Proprietary confidential information** 

© 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **TABLE OF CONTENTS** 1.

| TITLE PA | \GE1 |
|---|---|
| 1. | TABLE OF CONTENTS |
| LIST OF | TABLES4 |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY8 |
| 5.<br>5.1<br>5.2<br>5.2.1<br>5.2.2 | ENDPOINT(S) |
| 5.4.1 | Demographics and baseline characteristics9 |
| 6. | GENERAL ANALYSIS DEFINITIONS |
| 6.1 | TREATMENT(S) 11 |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS11 |
| 6.3 | SUBJECT SETS ANALYSED |
| 6.5 | POOLING OF CENTRES12 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS 12 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS |
| | PLANNED ANALYSIS |
| 7. | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS 14 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION |
| 7.3 | TREATMENT COMPLIANCE |
| 7.4 | PRIMARY ENDPOINT(S) |
| 7.4.1 | Primary analysis |
| 7.4.2 | Interim analysis |
| 7.5 | SECONDARY ENDPOINT(S) |
| 7.5.1 | Key secondary endpoint(s) |
| 7.5.2 | (Other) Secondary endpoint(s) |
| 7.7 | EXTENT OF EXPOSURE |
| 7.8 | SAFETY ANALYSIS |
| 7.8.1 | Adverse events 15 |
| 7.8.2 | Laboratory data |

| Proprietary co | onfidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| 7.8.3 | Vital signs |
| 7.8.4 | ECG |
| 7.8.5 | Others |
| 7.8.5.1 | PK parameters |
| 8. | REFERENCES 20 |
| 10. | HISTORY TABLE22 |
| IU. | |

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## LIST OF TABLES

| Table 6.2: 1 | Module A Important protocol deviations | 11 |
|---|---|---|
| Table 6.7: 1 | Nominal time points and windows for imaging | 12 |
| Table 6.7: 2 | Time windows for assignment of safety lab measurements to visits for | |
| | statistical analysis | 13 |
| Table 10: 1 | History table | 22 |

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

Include a list of all abbreviations used in the TSAP for Module A

| Term | Definition / description |
|--------|------------------------------------------------------------|
| AE | Adverse Event |
| BHM | Bayesian Hierarchical Model |
| CR | Complete Response |
| CTC | Common Terminology Criteria |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DC | Disease Control |
| DBL | Database Lock |
| DLT | Dose Limiting Toxicity |
| DM&SM | Boehringer Ingelheim Data Management and Statistics Manual |
| DoR | Duration of Response |
| DRA | Drug Regulatory Affairs |
| DMG | Dictionary Maintenance Group |
| ECOG | Eastern Cooperative Oncology Group |
| EMA | European Medicines Agency |
| FL | Follicular Lymphoma |
| ICH | International Conference on Harmonisation |
| IPD | Important Protocol Divations |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQRM | Medical Quality Review Meeting |
| MTD | Maximum Tolerated Dose |
| O*C | Oracle Clinical |
| OR | Objective Response |
| OS | Overall Survival |
| PD | Progression of Disease |
| PFS | Progression-Free Survival |
| PK | Pharmacokinetics |
| PR | Partial Response |
| PSTAT | Project Statistician |

# Boehringer Ingelheim TSAP for RI Trial No. 1381

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|--------|-----------------------------------------------|
| PT | Preferred Term |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| RECIST | Response Evaluation Criteria in Solid Tumours |
| REP | Residual Effect Period |
| RPM | Report Planning Meeting |
| SA | Statistical Analysis |
| SAE | Serious Adverse Event |
| SD | Stable Disease |
| StD | Standard Deviation |
| SMQ | Standardised MedDRA query |
| SOC | System Organ Class |
| TESS | Treatment Emergent Signs and Symptoms |
| ToC | Table of Contents |
| TMW | Trial Medical Writer |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |

#### 3. INTRODUCTION

As per ICH E9 [1], the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Master and Module A Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the Module A TSAP is based on the planned analysis specification as written in Master and Module A CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, Module A TSAP readers may consult the Master and Module A CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS® Version 9.4 or the latest version will be used for analyses.

R v3.5.1 and JAGS v4.3.0 or the latest versions will be used for BHM analysis.

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

Refer to the Master TSAP.

## 5. ENDPOINT(S)

## **5.1 PRIMARY ENDPOINT(S)**

Refer to the Master TSAP.

# 5.2 SECONDARY ENDPOINT(S)

## 5.2.1 Key secondary endpoint(s)

This section is not applicable because no key secondary endpoints have been defined in the CTP.

## **5.2.2** Secondary endpoint(s)

Refer to the Master TSAP.



#### 5.4.1 Demographics and baseline characteristics

Refer to the Master TSAP.



TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENT(S)

Patients in this Module of the clinical trial will receive BI 754111 combined with BI 754091 by i.v. infusion after signing the Master and Module A informed consent forms and completing the screening processes. Treatment will be administered every 3 weeks (1 cycle = 21 days).

For definition of treatment periods refer to the Master TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Table 6.2: 1 Module A Important protocol deviations

| | tegory<br>ode | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|---|
| A | | Entrance criteria not met | | | |
| | Ala | Inclusion criteria not met | | | |
| | Ala.1 | No measurable lesions according to RECIST 1.1 | Inclusion criterion (IN) 3 not met | None | Automatic |
| | A2a | Exclusion criteria met | | | |
| | A2a.1 | Previous treatment with an anti-LAG-3 agent. | Exclusion criterion (EX) 2 met | None | Automatic |

#### 6.3 SUBJECT SETS ANALYSED

#### Module A Screened Set:

This patient set includes all patients who have signed the informed consent for the study and module A. The screened set will be used for patient disposition tables.

#### Module A Treated Set (TS):

This patient set includes all patients who were documented to have received at least one dose of trial medications in Module A. The TS is used for both efficacy analysis and safety analyses.

#### Module A Pharmacokinetic Set (PKS):

This patient set includes all patients in the TS with at least one valid plasma concentration. PKS will be used for all pharmacokinetic analyses..



#### 6.5 POOLING OF CENTRES

This section is not applicable because centre/country is not included in the statistical analyses.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Refer to the Master TSAP.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Baseline values will be the measurements taken most recently prior to first administration of study drug in Module A.

Study day will be calculated relative to the date of the first administration of study drug in Module A. The day prior to first administration of study drug will be 'Day -1' and the day of first administration of study drug will be 'Day 1'; therefore 'Day 0' will not exist.

In order to identify whether consecutive imaging time points are missing for a given patient in this module, a nominal time point (i.e. Week 6, 12, 18 ... etc.) will be assigned to each and every image. This is achieved by creating windows for every radiological response assessment. These windows are defined in <u>Table 6.7: 1</u>.

Table 6.7: 1 Nominal time points and windows for imaging

| Nominal time point (weeks from start of study medication) | Due date of scans (days)* | Window (days) |
|---|---|---|
| 6 | 43 | 1 to ≤ 64 |
| 12 | 85 | 65 to ≤ 106 |
| 18 | 127 | $107 \text{ to} \le 148$ |
| 24 | 169 | 149 to $\leq$ 200 |
| 33 | 232 | 201 to ≤ 263 |
| 42 | 295 | 264 to ≤ 326 |
| 51 | 358 | 327 to ≤ 389 |
| Etc., 9 week interval | Etc. | Etc. |

<sup>\*</sup> The date of the first dose of study medication is Day 1

If a patient does not have an image in one of the windows described above, he/she will be said to have missed an assessment for that time point.

Table 6.7: 2 Time windows for assignment of safety lab measurements to visits for statistical analysis

| Window No. | Nominal visit | Nominal day | Interval |
|---|---|---|---|
| 0 | Cycle 1 | 1 | NA |
| 1 | Cycle 1 | 8 | [2,11] |
| 2 | Cycle 1 | 15 | [12,18] |
| 3 | Cycle 2 | 22 | [19,32] |
| 4 | Cycle 3 | 43 | [33,53] |
| n+1 | Cycle n | 21*(n-1)+1 | [21*(n-1)-9,<br>21*(n-1)+11] |
| 18 | EOT | 21*16+1 | [327, 351] |
| 19 | Safety Follow<br>up | 21*16+31 | [352, ∞] |

Note: n=3,4,5,...,16.

For patients discontinuing treatment before Cycle 16 or receive treatment beyond Cycle 16, identify the last treatment cycle n (>=3) and time windows of EOT and Safety Follow up will be:

| Window No. | Nominal visit | Nominal day | Interval |
|---|---|---|---|
| n+1 | Cycle n | 21*(n-1)+1 | [21*(n-1)-9,<br>21*(n-1)+11] |
| n+2 | ЕОТ | 21*n+1 | [21*n-9,<br>21*n+15] |
| n+3 | Safety Follow<br>up | 21*n+31 | [21*n+16, ∞] |

#### 7. PLANNED ANALYSIS

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Refer to the Master TSAP.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Refer to the Master TSAP.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for treatment compliance.

## 7.4 PRIMARY ENDPOINT(S)

#### 7.4.1 Primary analysis

Refer to the Master TSAP for BHM [2] approach description for the primary analysis of ORR.

For the BHM approach, a non-informative normal distribution with mean 0 and standard deviation of 2 is specified for the mean  $\mu$ . For the inter-cohort heterogeneity parameter  $\tau$ , a half normal distribution with parameter 1 is used which is a very conservative assumption regarding between-cohort variability and hence leads to only little borrowing of data across patient cohorts because there is little prior information on the strength of the correlation between the treatment effects across cohorts in Module A. The target response rate  $\tilde{p}_j$  of each cohort for the BHM approach are 20%, 20% and 10% respectively.

Prior to the primary analysis, the interim futility analysis is planned (section 7.4.2).

### 7.4.2 Interim analysis

An interim analysis was performed for each cohort in this Module per protocol. No decision was made based on the results as the recruitment had completed when the interim analysis was performed.

#### 7.5 SECONDARY ENDPOINT(S)

#### 7.5.1 Key secondary endpoint(s)

This section is not applicable because no key secondary endpoints have been defined in the CTP.

#### 7.5.2 (Other) Secondary endpoint(s)

Refer to the Master TSAP.



#### 7.7 EXTENT OF EXPOSURE

The numbers of cycle initiated will be summarized descriptively for each cohort.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set (TS). Analysis will be performed as defined in Section 7.3.4 of the CTP.

#### 7.8.1 Adverse events

Refer to the Master TSAP.

#### 7.8.2 Laboratory data

Refer to the Master TSAP.

## 7.8.3 Vital signs

N/A

#### 7.8.4 ECG

N/A

#### **7.8.5** Others

### 7.8.5.1 PK parameters

Actual sampling times will be listed. Raw concentration values will be summarized descriptively per time point. The derived PK parameters will be summarized descriptively.

As described in Section 5.3.1 of the Module A CTP, plasma concentration values will be used to support an exploratory model based analysis, using pooled data from other studies. These analyses will be done and reported outside of the CTR.



TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 8. REFERENCES

- 1. *CPMP/ICH/363/96:* "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version.
- 2. Berry SM, Broglio KR, Groshen S, Berry DA. Bayesian hierarchical modeling of patient subpopulations: Efficient designs of Phase II oncology clinical trial. Clinical Trials 10 (5), 720-734 (2013) [R18-2260].

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **HISTORY TABLE 10.**

History table Table 10: 1

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Initial | 02-NOV-20 | | None | This is the initial TSAP with necessary information for trial conduct |
| Final | 16-JUL-21 | | None | This is the final TSAP |
| Revised | 04-MAY-22 | | None | |



#### APPROVAL / SIGNATURE PAGE

Document Number: c38788170 Technical Version Number: 1.0

**Document Name:** 08-01-tsap-module-a-core1

**Title:** An open-label, Phase II trial evaluating the safety and efficacy of BI 754111 in combination with BI 754091 in in PD-(L)1 naïve and PD-(L)1 pretreated patient populations with advanced and/or metastatic solid tumours who have had at least one line of systemic therapy

## Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|--------------------------------|-----------|------------------------|
| Author | | 04 May 2022 17:10 CEST |
| Approval-Biostatistics | | 04 May 2022 17:13 CEST |
| Approval-Team Member Medicine | | 04 May 2022 19:02 CEST |
| Approval-Clinical Trial Leader | | 11 May 2022 12:01 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c38788170Technical Version Number:1.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|